CLINICAL TRIAL: NCT06666335
Title: A Prospective, Open-label, Single Arm, Multicenter, Post-authorization Efficacy and Safety Study of Subcutaneous Anakinra in Chinese Patients With Colchicine-resistant Familial Mediterranean Fever (FMF)
Brief Title: A Study to Evaluate Efficacy and Safety of Anakinra in Chinese Patients With Colchicine-resistent FMF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.ANAKIN-701
Record Dates: First submitted 2024-10-08; First posted 2024-10-30 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Familial Mediterranean Fever (FMF )
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anakinra (Experimental): Anakinra, once daily s.c. injection, starting dose of 100 mg/day for patients with body weight ≥ 50 kg and 1-2 mg/kg/day for patients with body weight < 50 kg for 6 months. For patients < 16 years and < 50 kg not responding sufficiently, the dose can be increased up to 4 mg/kg/day (max of 200 mg/day).
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Subcutaneous injections once daily for 6 months
  Other Names: Kineret

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of anakinra in Chinese patients with colchicine-resistand Familial Mediterranian Fever (FMF). The study consists of up to one month screening, to see if a patient is suitable to the study, 6 months of treatment with anakinra and one month safety follow up after last dose of anakinra. In total 3 patients, male and female from 2 years of age (minimum 10kg weight), will be enrolled to the study.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-arm, multi-center study, and this study consists of a 6-month treatment period with anakinra followed by a 4-Week period to evaluate safety of anakinra after the last dose of study drug i.e. at Month 7. The study is divided into three parts: screening, treatment period, and safety follow-up.

The patient will enter screening after informed consent is obtained and will undergo screening assessments to confirm eligibility. Duration of the screening period will be kept as short as possible and should not exceed 4 weeks.

Patients will be assigned to study drug after they have met all of the inclusion criteria and none of the exclusion criteria. Patients will receive daily subcutaneous treatment with anakinra for 6 months.

After the last dose of anakinra at Month 6, the safety will continue to be evaluated at a Safety Follow-up visit., at Month 7.

The primary endpoint will be change in the number of FMF attacks per month per patient from baseline to subsequent study visits, up to Month 6.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form signed by the patient or a legal guardian representative.
2. Male or female patients, 2 years of age or older with a body weight ≥ 10 kg.
3. Diagnosis of FMF confirmed by a positive genetic testing i.e., mutations in both alleles of the MEFV gene (i.e. homozygous or compound heterozygous).
4. Patient must have an estimated mean of at least 2 acute FMF attacks per month within 2 months prior to enrollment to the study.
5. Patient must be resistant to colchicine treatment.
6. Female patients of childbearing potential and male patients with female partners of childbearing potential must use an effective method of contraception during the study (abstinence being a possible option) as well as a negative pregnancy test prior to enrollment for females of childbearing potential and participating in the study.
7. Negative tuberculosis screening confirmed at screening visit by the Mantoux Tuberculin skin test (TST) using purified protein derivative (PPD), or by Interferon-Gamma-Release Assays (IGRAs) e.g., QuantiFERON® TB Gold Plus (QFT-Plus) or T-Spot® (TB Test) within 8 weeks prior to enrollment. Negative results must be complemented by the medical history, physical examination, and Chest X-Ray. Patients presenting positive TST or IGRA with or without active or clinical suspicion of latent tuberculosis are not eligible to enter the study. Previously vaccinated for Tuberculosis patients: IGRA positive patients are not eligible to enter the study; TST positive patients with an induration of 15 mm and more are also not eligible to enter the study, TST positive patients (with an induration up to 15 mm) are also not eligible to enter the study, unless an IGRA test is subsequently performed and provides a negative result.

Exclusion Criteria:

1. Previous enrollment to this study.
2. Participation in another clinical interventional study 30 days prior to enrollment.
3. Treatment with an investigational drug within 5 half-lives prior to enrollment.
4. Previous or current treatment with anakinra, or any other IL-1 inhibitor.

6. Live vaccines within 4 weeks prior to enrollment.

7. Known presence or suspicion of active, chronic or recurrent bacterial, fungal or viral infections, including but not limited to tuberculosis, HIV infection, Covid-19 infection, hepatitis B or C infection at baseline.

8. Clinical evidence of liver disease or liver injury as indicated by presence of abnormal liver tests

9. Presence of severe chronic kidney disease

10. Diagnosis of amyloidosis at baseline.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the number of FMF attacks per month. | Up to 6 Months
  An FMF attack is defined as fever ≥ 38°C lasting between 6 hours to 7 days and accompanied by painful serositis manifestations in any of the following sites: abdomen, chest, joints and skin.

SECONDARY OUTCOMES:
The number of months free of FMF attacks will be evaluated in each patient. | Up to 6 months.
  An FMF attack is defined as fever ≥ 38°C lasting between 6 hours to 7 days and accompanied by painful serositis manifestations in any of the following sites: abdomen, chest, joints and skin.
Change from baseline in C-reactive protein (CRP) concentrations. | Up to 6 months.
  CRP levels (measured in mg/L) will be determined in serum.
Change from baseline in Serum Amyloid A (SAA) concentrations. | Up to 6 months.
  SAA levels (measured in mg/L) will be determined in serum.
Change from baseline in the dose of analgesic agents used for the treatment of FMF symptoms. | Up to 6 months.
  Reduction in the dose (measured in mg/kg) of analgesic treatments for FMF attacks will be evaluated during the study.
Number of patients responding to study drug over time using the Modified FMF50 score. | Up to 6 months.
  Modified FMF50 score response is defined by the to the presence of 3 of the 4 following criteria: decrease by ≥ 50% in the frequency of all FMF attacks; decrease by ≥ 50% in the frequency of FMF attacks in the joints; decrease by ≥ 50% in the levels of either SAA or CRP (measured as mg/L) with target level concentrations for CRP and SAA ≤10 mg/L; Increase by ≥ 50% in QoL values assessed using the VAS scale (0-10cm), where scores of 0 and 10 indicate the lowest and highest QoL scores, respectively.
Number of Participants with Adverse Events (AEs), Serious Adverse Events (SAEs), deaths, and AEs leading to study drug discontinuation | Up to 7 months
  An AE is any untoward medical occurrence in a study patient to whom a medicinal product is administered, and which does not necessarily have a causal relationship with this treatment.
  AEs include abnormal test findings, clinically significant signs and symptoms, changes in physical examination findings, progression or worsening of underlying disease.
  Serious adverse events (SAEs) were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards.
Changes over time in vital signs | Up to 7 months
  Vital signs change of each patients are evaluated over time. The vital sign evaluated are blood pressure (mmHg), heart rate (beats per minute), and body temperature (Celsius degrees).
Changes over time in body weight and height | Up to 7 months
  Body weight (kilograms) and height (centimeters) of each patients are evaluated over time.
Changes over time in Laboratory safety assessment | Up to 7 months
  Number of patients with abnormal laboratory test results

IPD SHARING:
Plan to Share IPD: No